CLINICAL TRIAL: NCT04927546
Title: Impact of Interleukin-6 Receptor Blockade on Acute Response to Exercise on Insulin Sensitivity and Muscle Glucose Uptake in Patients With Rheumatoid Arthritis
Brief Title: Acute Response to Exercise in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IL-6 blockade and exercise
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RA patients will be divided into 2 groups, according to the pharmacological treatment (tocilizumab or anti-TNF). A third group will be composed by healthy controls. The acute responses of insulin sensitivity after an acute session of exercise will be assessed by the hyperinsulinemic euglycemic clamp, and the molecular pathways will be assessed by muscle biopsy and gene and protein expression analysis. Positron emission tomography-magnetic resonance imaging (PET/MRI) will be performed to quantify skeletal muscle glucose uptake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IL-6 blockade (Experimental): RA patients under pharmacological treatment with interleukin-6 blockade.
  Interventions: Behavioral: Exercise
- Anti-TNF-alpha (Experimental): RA patients under pharmacological treatment with anti-TNF-alpha.
  Interventions: Behavioral: Exercise
- Healthy controls (Experimental): Healthy participants.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Thirty minutes of aerobic exercise in a treadmill.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that affects the joints, causing pain, edema, physical disability and poor quality of life. In addition, RA patients are at increased risk of developing cardiovascular disease (CVD) and premature death. The most effective pharmacological treatment is the use of biological agents that inhibit the action of specific substances, such as interleukin 6 (IL-6) and tumor necrosis factors (TNF). Physical exercise is considered a first-line non-pharmacological treatment in RA, improving inflammatory and metabolic profile, functional capacity, fatigue and preventing the onset of CVD. There is evidence that IL-6, when secreted as a result of exercise, brings several benefits. However, there is no study investigating the interaction between biological IL-6 blocking agents and exercise on metabolic responses, such as insulin sensitivity and glucose uptake, in patients with RA. To answer this question, adult women diagnosed with RA and healthy controls will be recruited for an acute session of exercise. RA patients will be divided into 2 groups, according to the pharmacological treatment (tocilizumab or anti-TNF). The acute responses of insulin sensitivity after an acute session of exercise will be assessed by the hyperinsulinemic euglycemic clamp, and the molecular pathways will be assessed by muscle biopsy and gene and protein expression analysis. Positron emission tomography-magnetic resonance imaging (PET/MRI) will be performed to quantify skeletal muscle glucose uptake.

ELIGIBILITY:
Inclusion Criteria:

* Adult women diagnosed with rheumatoid arthritis under pharmacological treatment, for at least 6 months, with a monoclonal antibody against the interleukin-6 receptor or TNF-alpha inhibitors;
* Stable dose of monoclonal antibody against the interleukin-6 receptor or TNF-alpha inhibitors in the previous 3 months;

Exclusion Criteria:

* Any physical limitation or disability that preclude exercise participation;
* Participation in a structured exercise program in the previous 12 months;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 1 hour post-exercise
  Acute effect of exercise on insulin sensitivity assessed by the hyperinsulinemic euglycemic clamp.

SECONDARY OUTCOMES:
Insulin sensitivity-related molecular pathway (Western Blotting) | Baseline and 4 hours post-exercise
  Insulin sensitivity-related molecular pathway will be assessed by Western Blotting.
Insulin sensitivity-related molecular pathway (RT-PCR) | Baseline and 4 hours post-exercise
  Insulin sensitivity-related molecular pathway will be assessed by Real-Time Polymerase Chain Reaction (RT-PCR).
Skeletal muscle glucose uptake | 3 hours post-exercise
  Positron emission tomography-magnetic resonance imaging (PET/MRI) will be performed to quantify skeletal muscle glucose uptake.

CONTACTS AND LOCATIONS:
Locations (1):
- Univsersity of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casale AR, Lemes IR, Smaira FI, Astley C, Oliveira-Junior G, de Sa Pinto AL, de Medeiros-Ribeiro AC, Godoy-Santos AL, Lima M, Carneiro CG, Buchpiguel CA, Dantas WS, Axelrod CL, Javvadi P, Ghosh S, Kirwan JP, Roschel H, Gualano B. Interleukin-6 blockade does not impair exercise-induced glucose uptake and insulin sensitivity in rheumatoid arthritis. Am J Physiol Endocrinol Metab. 2025 Dec 1;329(6):E849-E860. doi: 10.1152/ajpendo.00348.2025. Epub 2025 Oct 17. PMID 41106846